CLINICAL TRIAL: NCT04753983
Title: fMRI of Active DBS Stimulation in Epilepsy
Brief Title: A Study to Evaluate fMRI of Active DBS Stimulation in Epilepsy
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No longer have funding
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Steven A. Messina, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 20-006464
Record Dates: First submitted 2021-02-09; First posted 2021-02-15 (Actual); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Refractory Epilepsy
Keywords: Deep Brain Stimulation
MeSH Terms: conditions — Drug Resistant Epilepsy | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Anterior Nucleus of the Thalamus (ANT) Deep Brain Stimulation (DBS) (Experimental): Subjects that have undergone DBS placement for treatment of refractory epilepsy will undergo a fMRI scan. During the fMRI, the subject will undergo alternating short periods of their DBS in the "on" and "off" state with high- and low frequency settings to measure the brain activation changes induced by the DBS.
  Interventions: Diagnostic Test: Functional magnetic resonance imaging (fMRI)

INTERVENTIONS:
Diagnostic Test: Functional magnetic resonance imaging (fMRI) — Diagnostic imaging measuring the metabolic changes that occur within the brain used for measuring and mapping brain activity

SUMMARY:
The purpose of this study is to use functional imaging to study the mechanisms of the anterior nucleus of the thalamus (ANT) deep brain stimulation (DBS).

DETAILED DESCRIPTION:
Researchers are testing how changing the settings on deep brain stimulation device (DBS) can help reduce the number and severity of seizures. Functional imaging will be used to study the mechanisms of ANT DBS to optimize the device settings to improve the degree of seizure reduction.

ELIGIBILITY:
Inclusion Criteria:

- Patients who have previously undergone anterior thalamic nucleus deep brain stimulation (DBS) for refractory epilepsy.

Exclusion Criteria:

- Contraindication to MRI; prior brain resective surgery or large area of brain tissue loss (e.g., large area infarction).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-09 (Estimated); Primary Completion 2024-05 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Document brain activation networks with ANT stimulation | Results would be available immediately following processing of the imaging data after each scan
  Use resting state fMRI to map brain network activation with high and low frequency of ANT stimulation.

CONTACTS AND LOCATIONS:
Overall Officials: Steven A Messina, MD, Principal Investigator — Mayo Clinic

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials